CLINICAL TRIAL: NCT01708304
Title: From Evidence-Base to Practice: Implementing RDAD in AAA Community-Based Services
Brief Title: Reducing Disabilities in Alzheimer's Disease (RDAD) Translation in Area Agencies on Aging (AAAs)
Acronym: RDAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Linda Teri, Professor, Psychosocial & Community Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41906
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer's Disease; Dementia; Memory Impairment; Cognitive Impairment
Keywords: Dementia; Alzheimer's Disease; Exercise; Caregiver; Behavior modification
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RDAD (Other): Exercise training for caregiver and care recipient. Behavior modification training for caregiver.
  Interventions: Behavioral: RDAD

INTERVENTIONS:
Behavioral: RDAD — Exercise training for caregiver and care recipient. Behavioral modification training for caregiver.

SUMMARY:
The University of Washington's Northwest Research Group on Aging is partnering with Area Agencies on Aging (AAA) in Washington and Oregon to complete this translational investigation of RDAD (Reducing Disabilities in Alzheimer's Disease). RDAD is an evidence-based program with demonstrated efficacy in helping older adults with dementia maintain physical function and remain physically and mentally healthy. This study asks two questions: 1) Can AAA partners successfully translate and implement RDAD, and 2) Is AAA implementation of RDAD effective in producing desired outcomes among agencies, providers, and older adults with dementia and their family members. This study is being conducted in Washington and Oregon states.

ELIGIBILITY:
Inclusion Criteria:

Care Recipients must

* Have a diagnosis of dementia
* Be 65 years of age or older
* Currently exercise no more than 150 minutes a week and not regularly participate in a formal exercise program.

Caregivers must

* Live in the community
* Provide care to the care recipient with dementia

Exclusion Criteria:

Either Care-recipient or Caregiver must not

* Plan to move to a long-term residential care setting within 6 months of enrollment.
* Plan to move from the study geographic area within 4 months of enrollment.
* Have a known terminal illness (with death anticipated within the next 12 months)
* Have had a hospitalization for a psychiatric disorder in the 12 months prior to baseline
* Be actively suicidal, hallucinating, or delusional
* Be blind, deaf, or not ambulatory

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 510 (Actual)
Dates: Start 2012-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Minutes of exercise per week | Change from baseline in number of minutes of exercise each week during treatment phase of study, weeks 7-12
  Caregivers will track the number of minutes per week the care recipients engage in exercise recommended by the coach.
Restricted Activity Days | Baseline
  Restricted Activity Days measures how much the participant cut down his/her usual activities in the previous two weeks because of injury or illness and how many days the participant stayed in bed in the previous two weeks because of injury or illness.
Restricted Activity Days | Change from Baseline to Pre-Treatment (6 weeks)
  Restricted Activity Days measures how much the participant cut down his/her usual activities in the previous two weeks because of injury or illness and how many days the participant stayed in bed in the previous two weeks because of injury or illness.
Restricted Activity Days | Change from Baseline to Post- Treatment 1 (13 weeks)
  Restricted Activity Days measures how much the participant cut down his/her usual activities in the previous two weeks because of injury or illness and how many days the participant stayed in bed in the previous two weeks because of injury or illness.
Restricted Activity Days | Change from Baseline to Post-Treatment 2 (30 weeks)
  Restricted Activity Days measures how much the participant cut down his/her usual activities in the previous two weeks because of injury or illness and how many days the participant stayed in bed in the previous two weeks because of injury or illness.
Restricted Days of Activity | Change from Baseline to 13 Month Follow-Up
  Restricted Activity Days measures how much the participant cut down his/her usual activities in the previous two weeks because of injury or illness and how many days the participant stayed in bed in the previous two weeks because of injury or illness.
Independence/Residential Status | Change from Baseline to 13 Month Follow-Up
  All participants will be in independent living situations at baseline. Any move from independent living to a care facility will be documented throughout the 13 month study.

SECONDARY OUTCOMES:
Revised Memory and Behavior Problem Checklist (RMBPC) | Baseline
  Checklist rates 24 care recipient behaviors for frequency of occurrence and caregiver reaction.
Revised Memory and Behavior Problem Checklist (RMBPC) | Change from Baseline to Pre-Treatment (6 weeks)
  Checklist rates 24 care recipient behaviors for frequency of occurrence and caregiver reaction.
Revised Memory and Behavior Problem Checklist (RMBPC) | Change from Baseline to Post-Treatment 1 (13 weeks)
  Checklist rates 24 care recipient behaviors for frequency of occurrence and caregiver reaction.
Revised Memory and Behavior Problem Checklist (RMBPC) | Change from Baseline to Post-Treatment 2 (30 weeks)
  Checklist rates 24 care recipient behaviors for frequency of occurrence and caregiver reaction.
Revised Memory and Behavior Problem Checklist (RMBPC) | Change from Baseline to 13 Month Follow-Up
  Checklist rates 24 care recipient behaviors for frequency of occurrence and caregiver reaction.
Quality of Life-AD | Baseline
  This 13-item measure is specifically designed for individuals with dementia and focuses on quality of life domains identified as important for cognitively impaired older adults.
Quality of Life-AD | Change from Baseline to Pre-Treatment (6 weeks)
  This 13-item measure is specifically designed for individuals with dementia and focuses on quality of life domains identified as important for cognitively impaired older adults.
Quality of Life-AD | Change from Baseline to Post-Treatment 1 (13 weeks)
  This 13-item measure is specifically designed for individuals with dementia and focuses on quality of life domains identified as important for cognitively impaired older adults.
Quality of Life-AD | Change from Baseline to Post-Treatment 2 (30 weeks)
  This 13-item measure is specifically designed for individuals with dementia and focuses on quality of life domains identified as important for cognitively impaired older adults.
Quality of Life-AD | Change from Baseline to 13 Month Follow-Up
  This 13-item measure is specifically designed for individuals with dementia and focuses on quality of life domains identified as important for cognitively impaired older adults.
CES-D | Baseline
  This 20-item scale that assesses depression in caregivers.
CES-D | Change from Baseline to Pre-Treatment (6 weeks)
  A 20-item scale that assesses depression in caregivers.
CES-D | Change from Baseline to Post-Treatment 1 (13 weeks)
  A 20-item scale that assesses depression in caregivers.
CES-D | Change from Baseline to Post-Treatment 2 (30 weeks)
  A 20-item scale that assesses depression in caregivers.
CES-D | Change from Baseline to 13 Month Follow-Up
  A 20-item scale that assesses depression in caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Teri, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Teri L, Logsdon RG, McCurry SM, Pike KC, McGough EL. Translating an Evidence-based Multicomponent Intervention for Older Adults With Dementia and Caregivers. Gerontologist. 2020 Apr 2;60(3):548-557. doi: 10.1093/geront/gny122. PMID 30304477